CLINICAL TRIAL: NCT01576887
Title: A Double-Blind, Randomized, Placebo-Controlled Safety Study Evaluating the Effects of Residual Renal Function (RFF) in Patients With End-Stage Renal Disease and Type 2 Diabetes Mellitus on Peritoneal Dialysis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-1201; 2012-001563-78 (EudraCT Number)
Record Dates: First submitted 2012-03-30; First posted 2012-04-13 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: End-Stage Renal Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus, Type 2 | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bardoxolone Methyl (Experimental)
  Interventions: Drug: Bardoxolone Methyl 20 mg

INTERVENTIONS:
Drug: Bardoxolone Methyl 20 mg — Oral, once daily
  Arms: Bardoxolone Methyl
Drug: Placebo — Oral, once daily
  Arms: Placebo

SUMMARY:
This study is a multi-center, double-blinded, randomized, study of bardoxolone methyl treatment in patients with End-Stage Renal Disease (ERSD) and Type 2 Diabetes Mellitus (T2DM) on peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have ESRD and been on PD for longer than 3 months
2. Patients must have had a diagnosis of T2DM prior to starting dialysis
3. Patients must have RRF, as defined by the mean of urea and creatinine clearance on a 24 hour urine collection, ≥ 25 Liters/week/1.73 m2 documented in the four months prior to the Screen A visit
4. Patients must have RRF, as defined by the mean of urea and creatinine clearances on a 24 hour urine collection, ≥ 25 Liters/week/1.73 m2 at both the Screen A and Screen B visits
5. The RRF value obtained at the Screen B visit, must not be less than 50% of the RRF value obtained at the Screen A visit
6. Patients must be at least 18 years of age
7. Patients must have a mean systolic blood pressure (SBP) on three readings at both Screen A and Screen B visits ≤ 160 mmHg and ≥ 90 mmHg
8. Patients must have a mean diastolic blood pressure (DBP) on three readings at both Screen A and Screen B visits < 100 mmHg and ≥ 40 mmHg
9. Patients must be willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested
10. Patients must be willing and able to cooperate with all aspects of the protocol
11. Patients must be willing and able to give written informed consent to participate in the study. They must provide consent for access to medical data according to appropriate local data protection legislation and allow authorization to access medical records that describe events captured in the endpoints

Exclusion Criteria:

1. History of Autosomal Dominant Polycystic Kidney Disease
2. Currently Active Systemic Lupus Erythematosus
3. History of Hepatitis B Surface Antigen +
4. History of Hepatitis C Antibody + being treated with antiviral therapy
5. History of an organ transplant
6. A planned renal transplant from a living donor during the study
7. History of hospitalization for congestive heart failure or pulmonary edema within 12 weeks before study randomization
8. History of cirrhosis of the liver
9. History of amyloidosis or light chain nephropathy
10. History of hemoglobin A1c level > 11.0% (97 mmol/mol) within 12 weeks before study randomization
11. History of recently active cardiovascular disease defined as:

    1. Unstable angina pectoris within 12 weeks before study randomization
    2. Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before study randomization
    3. Cerebrovascular accident, including transient ischemic attack within 12 weeks before study randomization
12. History of a diagnostic or interventional procedure that required intravenous administration of an iodinated contrast agent or gadolinium within 12 weeks before study randomization
13. History of known severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy
14. History of known 2o or 3o atrioventricular block not successfully treated with a pacemaker
15. History or resuscitated sudden cardiac death
16. History of an automatic implantable defibrillator
17. QTc greater than 0.50 seconds on an ECG obtained during either Screen A or Screen B visits
18. A serum magnesium level less than 1.4 meq/L on either Screen A or Screen B visit laboratory test results
19. History of systemic immunosuppression for more than 15 days, cumulatively, within the 12 weeks prior to study randomization or anticipated need for more than 15 days of immunosuppression during the study
20. Total bilirubin, aspartate transaminase (AST), or alanine transaminase (ALT) level greater than the upper limit of normal (ULN) or alkaline phosphatase level greater than two times the ULN on either the Screen A and Screen B visit laboratory test results
21. Known hypersensitivity to any component of the study drug
22. Current history of drug or alcohol abuse, as assessed by the investigator
23. History of clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 12 weeks before study randomization
24. In patients who have been on peritoneal dialysis for ≥ 6 months, two or more episodes of peritonitis in the 6 months before study randomization. In patients who have been on peritoneal dialysis for <6 months, one episode of peritonitis before study randomization
25. History of a diagnosis or treatment of a malignancy in the past 5 years, excluding non-melanoma skin cancer and carcinoma in situ of the cervix
26. History of a clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the patient while involved in the study
27. Patient is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
28. Participation in a clinical study involving any intervention within 30 days prior to Screen A visit, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form
29. Female patients who are pregnant, intend to become pregnant during this study, or are nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | Approximately 17 months

SECONDARY OUTCOMES:
Type of Adverse Events | Approximately 17 months
Change in Residual Renal Function | Baseline to 6 months
Maximum observed concentration | Day 0, 30, 60, 90, 120, 150, 180, 210
Time to maximum observed concentration | Day 0, 30, 60, 90, 120, 150, 180, 210
Area under the plasma concentration-time curve | 2, 4, 8, 24 hours, 30, 60, 90, 120, 150 and 180 days
  Only the first 8 patients randomized will have the PK drawn and hours 2, 4, 8, and 24. All patients will have the PK drawn at 30, 60, 90, 120, 150 and 180 days.
Area under the curve | 2, 4, 8 and 24 hours
  Only the first 8 patients randomized

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/